CLINICAL TRIAL: NCT01584388
Title: Rituximab (RTX) for IgG4-related Disease (IgG4-RD): a Prospective,Open-label Trial
Brief Title: Rituximab in IgG4-RD: A Phase 1-2 Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, John H. Stone, MD, Director, Clinical Rheumatology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011p002414
Record Dates: First submitted 2012-04-22; First posted 2012-04-25 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Retroperitoneal Fibrosis; Autoimmune Pancreatitis; Sialadenitis; Pseudotumor
Keywords: Type 1 autoimmune pancreatitis; IgG4-related sclerosing cholangitis; Chronic sclerosing sialadenitis; Lacrimal glands; Orbital pseudotumor; IgG4-related tubulointerstitial nephritis; Lymphadenopathy; Pachymeningitis; Aorta; Peri-aortitis; Retroperitoneal fibrosis; Riedel's thyroiditis
MeSH Terms: conditions — Retroperitoneal Fibrosis; Autoimmune Pancreatitis; Sialadenitis; Orbital Pseudotumor; Lymphadenopathy; Meningitis | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab 1000 mg IV times two doses, separated by approximately 15 days.
  Other Names: Rituxan

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of rituximab in IgG4-RD.

DETAILED DESCRIPTION:
This two-center trial will enroll at total of 30 patients with IgG4-RD. The two participating sites are the Massachusetts General Hospital (Boston, MA) and the Mayo Clinic (Rochester, MN). All patients will receive rituximab 1 gram intravenously times two doses, separated by approximately 15 days. The primary efficacy outcome - disease remission and successful completion of the glucocorticoid taper - will be assessed at six months. Patients will be followed on the protocol for an additional six months after measurement of the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the trial based on the following disease-specific criteria:

* Age 18 or older
* Diagnosis of IgG4-RD, based upon either pathological criteria* (for those who have undergone biopsies) or clinical criteria.** The criteria for pathological and clinical diagnoses are specified below.

  * The subject can be either steroid-naive, in relapse, steroid dependent, or refractory to steroids. Subjects who are steroid dependent or refractory are eligible for enrollment if steroid dose has not been increased in the past 2 weeks, and their treating physician plans to withdraw steroids completely (by dose taper) within 8 weeks of starting rituximab.

    * Pathological diagnosis:

      * Histopathologic features consisting of a lymphoplasmacytic infiltrate and storiform fibrosis within involved organs. Other histopathologic features consistent with IgG4-RD (e.g., obliterative phlebitis) may be present but are not required.
      * Either an IgG4/IgG plasma cell ratio of > 50% within the affected organs or more than 10 IgG4-bearing plasma cells per high-power field.

All patients with pathologic diagnoses will have their specimens reviewed by pathology investigators.

**Clinical diagnosis:

• Organ involvement in a pattern consistent with IgG4-RD. This must include dysfunction of one of the following organs: pancreas (autoimmune pancreatitis); salivary glands (chronic sclerosing sialadenitis); lacrimal glands; orbital pseudotumor; kidneys; lungs; lymph nodes; meninges; aorta (including aortitis/periaortitis and/or retroperitoneal fibrosis); thyroid gland (Riedel's thyroiditis). If a patient is enrolled with a clinical diagnosis alone, the diagnosis must be accompanied by both an imaging finding compatible with IgG4-RD and a 1.5-fold elevation in the serum IgG4 concentration.

Exclusion Criteria:

Patients will be excluded from the study based on the following criteria:

Disease-Specific Concerns: Excessive fibrosis within organs, such that a disease response to rituximab would not be expected.

General Medical Concerns:

* Pregnancy (a negative serum pregnancy test should be performed for all women of childbearing potential within 7 days of treatment), or lactating.
* Inability to comply with study and/or follow-up procedures.

Rituximab-Specific Concerns:

* History of HIV.
* Presence of active infection.
* New York Heart Association Classification III or IV heart disease (See Appendix D).
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* At the Investigator's discretion, receipt of a live vaccine within 4 weeks prior to randomization.
* Positive hepatitis B or C serology is considered a potential exclusion criterion. Hepatitis B screening should include hepatitis B antibody and surface antigen for a patient with no risk factors. For patients with risk factors or previous history of hepatitis B, add core antibodies and e-antigen.
* Allergies: History of severe allergic reactions to human or chimeric monoclonal antibodies or murine protein.
* Uncontrolled disease: They show evidence of other uncontrolled disease, including drug and alcohol abuse, which that could interfere with participation in the trial according to the protocol.
* History of anti-human anti-chimeric antibody formation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H Stone, MD, MPH, Study Chair — Massachusetts General Hospital (Rheumatology Unit); Arezou Khosroshahi, MD, Study Director — Massachusetts General Hospital (Rheumatology Unit)

REFERENCES:
- [Derived] Carruthers MN, Topazian MD, Khosroshahi A, Witzig TE, Wallace ZS, Hart PA, Deshpande V, Smyrk TC, Chari S, Stone JH. Rituximab for IgG4-related disease: a prospective, open-label trial. Ann Rheum Dis. 2015 Jun;74(6):1171-7. doi: 10.1136/annrheumdis-2014-206605. Epub 2015 Feb 9. PMID 25667206

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Covient sample
Arm/Group | Rituximab
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: IgG4-RD RI Score at Baseline and Six Months After Rituxan Treatment
Description: The IgG4-RD RI is then calculated by adding the individual organ scores.At each assessment, the physician enters a 0-4 score after the organ/site listed with:
  0 = Normal or resolved
  1. = Improved but still present
  2. = Persistent (still active; unchanged from previous visit)
  3. = New or recurrent disease activity while patient is off treatment
  4. = Worsened or new disease despite treatment Definitions Organ/Site score: The overall level of IgG4-RD activity within a specific organ system Symptomatic: Is the disease manifestation in a particular organ system symptomatic? (Y = yes; N = no) Urgent disease: Disease that requires treatment immediately to prevent serious organ dysfunction (Y = yes; N = no) (Presence of urgent disease within an organ leads to DOUBLING of that organ system score) Damage: Organ dysfunction that has occurred as a result of IgG4-RD and is considered permanent (Y = yes; N = no)
  The Responder Index ranges from 0-60.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- IgG4-RD Responder Index: Scoring at baseline
- 6 Months: IgG4-RD Responder Index 6 months after treatment
Arm/Group | IgG4-RD Responder Index | 6 Months
Number analyzed (Participants) | 30 | 30
units on a scale | 11 (7) | 1 (2)

2. Primary Outcome: Cumulative Glucocorticoid Use at Baseline and 6 Months
Description: Cumulative glucocorticoid therapy between baseline and 6 months.
Time Frame: 6 months
Population: cumulative glucocorticoid use at 6 and compare them to baseline using paired T tests.
Measure: Mean (Full Range); unit: mg
Groups:
- Glucocorticoid Treatment (Baseline): total prednisone dose equivalent (mg) admin in the 28 preceding enrollment)
- Glucocorticoid Use (6 Months): total prednisone dose equivalent admin over 28 days prior to the 6 month study visit
Arm/Group | Glucocorticoid Treatment (Baseline) | Glucocorticoid Use (6 Months)
Number analyzed (Participants) | 30 | 30
mg | 42 [0 to 850] | 15 [0 to 280]

3. Primary Outcome: No Disease Flares During Rituximab Treatment Phase
Description: Disease flare measured by responder Index score:
  At each assessment, the physician enters a 0-4 score after the organ/site listed with:
  0 = Normal or resolved
  1. = Improved but still present
  2. = Persistent (still active; unchanged from previous visit)
  3. = New or recurrent disease activity while patient is off treatment
  4. = Worsened or new disease despite treatment Definitions Organ/Site score: The overall level of IgG4-RD activity within a specific organ system Symptomatic: Is the disease manifestation in a particular organ system symptomatic? (Y = yes; N = no) Urgent disease: Disease that requires treatment immediately to prevent serious organ dysfunction (Y = yes; N = no) (Presence of urgent disease within an organ leads to DOUBLING of that organ system score) Damage: Organ dysfunction that has occurred as a result of IgG4-RD and is considered permanent (Y = yes; N = no)
Time Frame: Month 6
Population: number of subjects without disease flares during baseline to 6 month of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Disease Flare: no disease flare before month 6
Arm/Group | Disease Flare
Number analyzed (Participants) | 30
Participants | 23

4. Secondary Outcome: Retreatment With Rituximab for Disease Relapse
Description: Number of subjects that relapsed during the course of the trial
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Relapse Treatment: Rituximab treatment for relapse
Arm/Group | Relapse Treatment
Number analyzed (Participants) | 30
Participants | 4

5. Secondary Outcome: Disease Response at 6 Months
Description: Decline of IgG4-RD Responder Index by at least two points for at least 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Disease Response at 6 Months: Decline of IgG4-RD RI by at least 2 points and maintained at 6 months.
Arm/Group | Disease Response at 6 Months
Number analyzed (Participants) | 30
Participants | 29

6. Secondary Outcome: Sustained Disease Response
Description: Decline of the IgG4-RD RI by at least two points and maintained for 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Disease Response at 12 Months: Decline of IgG4-RD RI by at least 2 points and maintained at 12 months.
Arm/Group | Disease Response at 12 Months
Number analyzed (Participants) | 30
Participants | 22

7. Secondary Outcome: Complete Remission
Description: IgG4-RD RI (including serum IgG4) of 0 at six months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Complete Remission at 6 Months: IgG-RD RI (exclusive of serum IgG4) of 0 at 6 months.
Arm/Group | Complete Remission at 6 Months
Number analyzed (Participants) | 30
Participants | 14

8. Secondary Outcome: Complete Remission IgG-RD RI (Exclusive of Serum IgG4) of 0 at 6 Months.
Description: IgG-RD RI (exclusive of serum IgG4) of 0 at 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Complete Remission at 6 Months, Exclusive of Serum IgG4: IgG-RD RI (exclusive of serum IgG4) of 0 at 6 months.
Arm/Group | Complete Remission at 6 Months, Exclusive of Serum IgG4
Number analyzed (Participants) | 30
Participants | 18

9. Secondary Outcome: Complete Remission at Any Timepoint
Description: IgG4-RD RI = 0 at any point in the trial
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Complete Remission (Any Timepoint): IgG4-RD RI = 0 at any point in the trial
Arm/Group | Complete Remission (Any Timepoint)
Number analyzed (Participants) | 30
Participants | 18

10. Secondary Outcome: Complete Remission (Any Timepoint), Exclusive of Serum IgG4
Description: IgG4-RD RI = 0 (exclusive of serum IgG4) at any point in the trial
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Complete Remission at Any Timepoint, Exclusive of Serum IgG4: IgG4-RD RI = 0 (exclusive of serum IgG4) at any point in the trial
Arm/Group | Complete Remission at Any Timepoint, Exclusive of Serum IgG4
Number analyzed (Participants) | 30
Participants | 20

11. Secondary Outcome: Time to Disease Response
Description: Treatment phase up to 52 weeks (365 days)
Time Frame: Mean days +/- standard deviation
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Time to Disease Response: Time to achievement of IgG4-RD RI improvement of > 2
Arm/Group | Time to Disease Response
Number analyzed (Participants) | 30
Days | 43 (37)

12. Secondary Outcome: Time to Relapse
Description: Treatment phase up to 52 weeks (365 days)
Time Frame: Days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Time to Relapse: Time to increase in IgG4-RD RI and reinstitution of treatment
Arm/Group | Time to Relapse
Number analyzed (Participants) | 30
Days | 210 (105)

13. Secondary Outcome: Time to Complete Remission
Description: Treatment phase up to 52 weeks (365 days)
Time Frame: Days
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Time to Complete Remission: Time to achievement of IgG4-RD RI of 0
Arm/Group | Time to Complete Remission
Number analyzed (Participants) | 30
Days | 198 (87)

ADVERSE EVENTS:
Time Frame: Reports of unanticipated problems involving risks to subjects or others are within 5 working days/7 calendar days of the date the investigator first becomes aware of the problem.
Description: Serious adverse event means any event temporally associated with the subject's participation in research that meets any of the following criteria:requires inpatient hospitalization or prolongation of existing hospitalization;
Groups:
- Open Label Treatment With Rituximab: Rituximab 1000 mg IV times two doses, separated by approximately 15 days
Arm/Group | Open Label Treatment With Rituximab
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment With Rituximab (N=30)
Legionella pneumophila pneumonia (Infections and infestations) | 1 (1) — The Legionella infection was present unrecognised at the time of the baseline infusion
Klebsiella urinary tract infection (Infections and infestations) | 1 (1) — Infection
cold agglutininmediated (Blood and lymphatic system disorders) | 1 (1)
Amaurosis fugax (Vascular disorders) | 1 (1) — amaurosis fugax leading to a carotid endarterectomy
unstable angina (Cardiac disorders) | 1 (1)
Surgery for pseudotumor (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No